CLINICAL TRIAL: NCT03278795
Title: Volume Support Ventilation Versus Pressure Support Ventilation as a Weaning Mode of Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Brief Title: VSV Versus PSV as a Weaning Mode of Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Taghyan, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VSVVPSVAAWMOMVCOPDP
Record Dates: First submitted 2017-08-25; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: COPD
Keywords: Weaning, ventilatory support, assisted ventilation modes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study group will be assigned to SIMV-VC for at least 48 hours . Patients will be assessed daily for fulfillment of criteria of readiness to wean according to European Respiratory Society guidelines (ERS guidelines ).
  After fulfillment of ERS weaning criteria patients will be consequently divided into two equal groups: 1. 25 patients will be assigned to PSV weaning mode.
  2. 25 patients will be assigned to VSV weaning mode. In PSV weaning group , PS will be adjusted 8 cm H2O. In VSV weaning group ,VT will be adjusted 6 ml/ Kg. Extubation will be done after successful spontaneous breathing trial according to ERS guidelines .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSV mode (Active Comparator): PSV weaning group
  Interventions: Procedure: pressure support ventilation mode
- VSV mode (Experimental): VSV weaning group
  Interventions: Procedure: volume support ventilation mode

INTERVENTIONS:
Procedure: pressure support ventilation mode — PSV is the sole mode of mechanical ventilation and will be used as a weaning mode in mechanically ventilated chronic obstructive pulmonary disease patients,In PSV weaning group , PS(pressure support) will be adjusted at 8 cmH2O until 2-h successful spontaneous breathing trial parameters according to ERS(European Respiratory Society) guidelines will be achieved and then patient will ex-tubated.
  Arms: PSV mode
Procedure: volume support ventilation mode — VSV mode could be viewed as "PRVC for spontaneous breathing" as it delivers a variable pressure to meet a target VT. VSV will be used as a weaning mode in mechanically ventilated chronic obstructive pulmonary disease patients,In VSV weaning group ,VT(tidal volume ) will be adjusted at 6 ml/ Kg until 2-h successful spontaneous breathing trial parameters according to ERS guidelines will be achieved and then patient will ex-tubated.
  Arms: VSV mode

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases. Acute exacerbations may occur during the management of stable COPD which can negatively impact health status, rates of hospitalization and re-admission. During exacerbation, some patients need immediate admission to the respiratory intensive care unit (RICU) for ventilatory support. As prolonged mechanical ventilation has unfavourable impacts, it is Important to minimize the duration of mechanical ventilation and perform extubation as soon as possible. In recent years, development of numerous models of artificial respiration, which could support spontaneous breathing, has made it possible to gradually decrease the mechanical ventilatory support. From these new modes, PSV which is a well known weaning mode will be compared in our study to a new weaning mode which is a volume support ventilation (VSV).

DETAILED DESCRIPTION:
Acute exacerbations may occur during the management of stable COPD which can negatively impact health status, rates of hospitalization and re-admission. During exacerbation, some patients need immediate admission to the respiratory intensive care unit (RICU). Ventilatory support in an exacerbation can be provided by either noninvasive (nasal or facial mask) or invasive (oro-tracheal tube or tracheostomy) ventilation.

Mechanical ventilation may be complicated by barotrauma, volutrauma, and also unfavourable impacts on cardiovascular system and organ perfusion. Moreover, prolonged mechanical ventilation enhances the risk of nosocomial pneumonia. So it is Important to minimize the duration of mechanical ventilation and perform extubation as soon as possible. In recent years, development of numerous models of artificial respiration, which could support spontaneous breathing, has made it possible to gradually decrease the mechanical ventilatory support.

From these new modes, PSV (pressure-support ventilation) which is a well known weaning mode will be compared in our study to a new weaning mode which is a volume support ventilation (VSV).

VSV could be viewed as "PRVC for spontaneous breathing" as it delivers a variable pressure to meet a target VT.

* The ventilator gives a test breath with an inspiratory pressure of 10 cmH2O above PEEP (5 cmH2O in earlier software versions)
* It measures the volume delivered and calculates system Compliance
* For each subsequent breath, the ventilator calculates compliance of the previous breath and adjusts the inspiratory pressure level (pressure level) to achieve the set VT on the next breath
* The ventilator will not change the inspiratory pressure by more than 3 cm H2O from one breath to the next
* Maximum available inspiratory pressure level is 5 cm H2O below the preset upper pressure limit (alarm will sound at this point and the breath will switch into exhalation)
* The minimum pressure limit is the baseline setting (PEEP)
* If apnea occurs, back up pressure control is activated and an alarm sounds
* If Auto mode is on and patient becomes apneic, the mode will automatically switch to PRVC(pressure regulated volume control).

In PSV patients in whom a 8 cm H2O pressure support level could be achieved,a 2-h trial of spontaneous breathing with this pressure support level will performed before extubation .

In the VSV group, VT(tidal volume) will be adjusted at 6 ml/ Kg and If the patients showed good tolerance with an acceptable ABG (arterial blood gas)analysis (pH o7.35, PaO2(partial pressure of arterial oxygen)/FIO2 .150 with an FIO2(fraction of inspired oxygen) f 40%, RR (respiratory rate) f 35 breaths/min), they will ventilated for 2-h trial of spontaneous breathing and then extubated

ELIGIBILITY:
Inclusion Criteria:

* All mechanically ventilated COPD patients at RICU.

Exclusion Criteria:

* COPD patients associated bronchiectasis , interstitial lung disease and pneumonia.
* Neurological and neuromuscular diseases hindering the respiratory drive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Success rate | the first 48 hours after ex-tubation from mechanical ventilation .
  Assess success rate of PSV and VSV in weaning of COPD patients .Weaning success is defined as extubation and the absence of ventilatory support 48h following the extubation .

SECONDARY OUTCOMES:
Detection of response to both modes | the first 48 hours after ex-tubation from mechanical ventilation .
  if there was a decrease in the total weaning time ,assisted ventilation time and total time of mechanical ventilation .
Number of weaning trials | the first 48 hours after ex-tubation from mechanical ventilation .
  Detection of number of spontaneous breathing trials needed for weaning among both modes

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes PJ, Celli BR. Systemic manifestations and comorbidities of COPD. Eur Respir J. 2009 May;33(5):1165-85. doi: 10.1183/09031936.00128008. PMID 19407051
- [Background] Sancar NK, Ozcan PE, Senturk E, Selek C, Cakar N. The Comparison of Pressure (PSV) and Volume Support Ventilation (VSV) as a 'Weaning' Mode. Turk J Anaesthesiol Reanim. 2014 Aug;42(4):170-5. doi: 10.5152/TJAR.2014.61687. Epub 2014 May 29. PMID 27366416
- [Background] Ruiz-Santana S, Garcia Jimenez A, Esteban A, Guerra L, Alvarez B, Corcia S, Gudin J, Martinez A, Quintana E, Armengol S, et al. ICU pneumonias: a multi-institutional study. Crit Care Med. 1987 Oct;15(10):930-2. doi: 10.1097/00003246-198710000-00007. PMID 3652708
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624